CLINICAL TRIAL: NCT06682390
Title: Contribution of Race to Nutritional Approach to Lower Cardiovascular Risk Factors in Men Undergoing Androgen Deprivation Therapy
Brief Title: Role of Race in Nutritional Approach in Men on ADT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Zhaoping Li, UCLA Professor of Medicine, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-001730
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer Metastatic Disease
Keywords: ADT; cardiovascular risk factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual dietary and physical activity regimen (No Intervention): Participants will maintain their habitual dietary and physical activity regimen for the first 3 months of the study.
- Hypocaloric anti-inflammatory diet (Experimental): Participants will follow a hypocaloric anti-inflammatory diet for the last 3 months of the study.
  Interventions: Behavioral: Hypocaloric anti-inflammatory diet

INTERVENTIONS:
Behavioral: Hypocaloric anti-inflammatory diet — The anti-inflammatory hypocaloric diet combines the exclusion of pro- inflammatory constituents and inclusion of anti-inflammatory nutrients. Excluded food items will be refined carbohydrates, soda and alcoholic beverages, ultra- processed foods, smoked foods, fatty foods, packaged foods, canned products, preservatives, emulsifiers, and sauces. Reduce or eliminate red/processed meats. Included food items will be a defined minimum diversity of fruits, vegetables, and nuts based on complementary phytonutrient contents, particularly those rich in phenolic compounds such as ellagitannins and sulforaphanes. Selected herbs (e.g., turmeric, ginger, garlic, black pepper, rosemary, cardamon, cinnamon), green tea, fermented foods, fats (e.g., avocado), and oils (e.g., olive oil) will be encouraged. The goal is to have 5 servings of vegetables, 2 fruits per day, and 5 vegetable color groups per week. Participants will also be asked to reduce their kcal by 500/day and walk for 1 gr 3x per week.
  Arms: Hypocaloric anti-inflammatory diet

SUMMARY:
There is a well-documented association between androgen deprivation therapy (ADT) and cardiovascular morbidity. A majority of men on ADT gain weight contributing to an increase in cardiovascular risk factors (CVRFs) and cardiovascular morbidity. Dietary intervention combined with exercise have shown success in reducing weight/fat mass and improving cardiovascular risk factors (CVRF). There is little data on whether African American men would respond to diet and exercise interventions differently from non-Hispanic white men. We will conduct a pilot, controlled two-phase intervention study stratified by race to investigate the following objectives:

1. Compare effect of a hypocaloric, anti-inflammatory diet on changes in fat mass between African- American vs non-Hispanic white men with metastatic prostate cancer on ADT therapy.
2. Compare effect of a hypocaloric, anti-inflammatory diet on changes in cardiovascular risk factors (body weight, lean body mass, waist-to-height ratio, blood pressure, lipids and HbA1C) and inflammatory markers (hs-CRP and cytokines) between African-American vs non-Hispanic white men with metastatic prostate cancer on ADT therapy.
3. Compare effect of a hypocaloric, anti-inflammatory diet on changes in cancer-related fatigue and quality of life between African-American vs non-Hispanic white men with metastatic prostate cancer on ADT therapy.

We will enroll 35 African American and 35 non-Hispanic white men with prostate cancer undergoing ADT therapy. In phase 1, after baseline assessment, men will consume their habitual diet and continue their habitual activity level for 3 months. During phase 2, participants will be instructed to consume a hypocaloric (-500 kcal), anti- inflammatory diet and walk for 1 hour on 3 days per week for 3 months. At baseline, after phase 1 and 2 primary outcome (fat mass) and secondary outcomes (CVRF and inflammatory markers) and tertiary outcomes (cancer-related fatigue and quality of life) will be determined.

ELIGIBILITY:
Inclusion Criteria:

* >12 months on ADT
* Expected continuation of ADT for >6 months upon initiation of study procedures
* Serum testosterone <50 ng/dL
* BMI >25
* Age >18 years old
* African American and Non-Hispanic white males
* Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent

Exclusion Criteria:

* Life expectancy < 1 year
* Females
* Radiation or chemotherapy treatment
* History of diabetes or serious medical condition including uncontrolled hypertension, liver, kidney, and cardiovascular disease
* Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator
* Any subject who currently uses tobacco products
* Any use of >20 g of alcohol per day
* Any subject who is unable or unwilling to comply with the study protocol
* Any subject who is unable to provide consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-11-20 (Estimated); Study Completion 2027-11-29 (Estimated)

PRIMARY OUTCOMES:
Fat mass | At baseline, 3 months and 6 months
  Bioelectric impedance measurement will provide information about body composition including percent body fat, fat mass, lean body mass, total body water and basal metabolic rate using the portable BIA310e (Biodynamics Corp.). BIA is based on the principle that the flow of an electrical current through an object can be used to determine the object's physical properties.
Waist circumference | At baseline, 3 months and 6 months
  Waist circumference will be measured with a tape measure in standing position horizontally, just above the hip bone, without compressing the skin.

SECONDARY OUTCOMES:
Blood lipids and lipoproteins (triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol) | At baseline, 3 months and 6 months
  Blood lipids and lipoproteins will be analyzed spectrophotometrically using reagent from Pointe Scientific (Canton, MI, USA).
HbA1c | At baseline, 3 months and 6 months
  HbA1c will be analyzed spectrophotometrically using reagent from Pointe Scientific (Canton, MI, USA).
Total testosterone | At baseline, 3 months and 6 months
  Total testosterone will be analyzed spectrophotometrically using reagent from Pointe Scientific (Canton, MI, USA).
Inflammatory markers (hs-CRP, IL-6, IL-1b, TNFa) | At baseline, 3 months and 6 months
  Concentrations of hs-CRP and cytokines will be quantified using the MagPix® analyzer (Luminex, Austin TX) with MILLIPLEX MAP Human CVD Panel 3 kit (hs-CRP) and Milliplex Human Cytokine/Chemokine MAGNETIC BEAD kit (IL-6, IL-1β, TNFα,) from EMD Millipore (Billerica, MA) at the Center for Human Nutrition Biomarker Laboratory.
Serum free fatty acids | At baseline, 3 months and 6 months
  Serum free fatty acids will be measured using an enzymatic colorimetric assay according to manufacturer (Sigma-Aldrich, St. Louis, MI).
Diet and physical activity | At baseline, 3 months and 6 months
  Participants in both groups will be instructed to use the weekly checklist for logging intake, physical activity and sleep habits. Subjects will be encouraged to track dietary intake as often as possible and mandated to complete 3-day dietary record 2 times every 4 weeks. Activity/exercise and sleep time will be monitored by the provided weekly checklist and ASA-24 at baseline, month 3, and month 6.

OTHER OUTCOMES:
Cancer-related fatigue | At baseline, 3 months and 6 months
  Participants will be asked to fill out a questionnaire about cancer-related fatigue.
Quality of life | At baseline, 3 months and 6 months
  Participants will be asked to fill out a questionnaire about quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles; Matthew Rettig, MD, Principal Investigator — Greater Los Angeles Division of Veterans Affairs, Los Angeles, California 90073
Locations (2):
- United States (2):
  - Greater Los Angeles Division of Veterans Affairs, Los Angeles, California
  - UCLA Health 200 Medical Plaza, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No